CLINICAL TRIAL: NCT01016509
Title: Tight Glycemic Control During Angioplasty Revascularization for Acute Coronary Syndrome Reduces Circulating Inflammatory Cytokines and Coronary Stent Restenosis
Brief Title: Tight Glycemic Control During Angioplasty Revascularization Reduces Coronary Stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, Assistant Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT 246813
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Restenosis; Tight Glycemic Control
Keywords: restenosis; insulin; hyperglycemia
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): No hyperglycemia patient group
- Insulin 1 (Active Comparator): Conventional insulin treatment
  Interventions: Drug: Insulin
- Insulin (Experimental): Intensive insulin treatment
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin infusion will be started when blood glucose levels exceeded 140 mg/dl and adjusted to maintain glycemia at 80-140 mg/dl. During insulin infusion, oral feeding will be stopped and parenteral nutrition (13±5 Kcal/kg-1/day-1) will be started. After the start of insulin infusion protocol a glycemic control will be provided every hour in order to obtain three consecutive values that were within the goal range. The infusion will be lasted until stable glycemic goal (80-140 mg/dl) at least for 24 h. After glycemic goal will be maintained for 24 h, a parenteral nutrition was stopped and feeding will be started according to European guidelines. Subcutaneous insulin will be initiated at the cessation of the infusion. After discharge from the hospital, insulin will be given as short-acting insulin before meals and long-acting insulin in the evening for 30 days from PCI. The treatment goal will be a fasting blood glucose level of 90-140 mg/dl and a non-fasting level of <180 mg/dl.
  Arms: Insulin
Drug: Insulin — Continuous insulin infusion of 50 IU Actrapid HM (Novo Nordisk) in 50 ml NaCl (0.9% using a Perfusor-FM pump) will be started only when blood glucose levels exceeded 200 mg/dl and adjusted to keep blood glucose between 180 and 200 mg/dl. When blood glucose fell <180 mg/dl, insulin infusion will be tapered and eventually stopped.The infusion will be lasted until stable glycemic goal (180-200 mg/dl) at least for 24 h. After glycemic goal will be maintained for 24 h, a parenteral nutrition was stopped and feeding will be started according to European guidelines. Subcutaneous insulin will be initiated at the cessation of the infusion. After discharge from the hospital, insulin will be given as short-acting insulin before meals and long-acting insulin in the evening for 30 days from PCI in both group. The treatment goal will be fasting blood glucose and postprandial levels of <200 mg/dl.
  Arms: Insulin 1

SUMMARY:
A multicentric study will evaluate whether peri-procedural tight glycemic control during angioplasty revascularization for acute coronary syndrome (ACS) reduces circulating inflammatory cytokines and thrombus formation in hyperglycaemic patients. Moreover, the investigators will assess whether the tight glycemic control during the first month from coronary event reduces the incidence of coronary stent restenosis at 6-months from PCI.

DETAILED DESCRIPTION:
The study design will be structured on the basis of protocol Yale. Upon emergency wards admission, all patients will be assigned to undergo prompt coronary revascularization. After PCI procedures, hyperglycemic patients will be randomly assigned to intensive glucose control (IGC group) and those treated with conventional glucose control (CGC group). In the patients with In the CGC group, continuous insulin infusion of 50 IU Actrapid HM (Novo Nordisk) in 50 ml NaCl (0.9% using a Perfusor-FM pump) will be started only when blood glucose levels exceeded 200 mg/dl and adjusted to keep blood glucose between 180 and 200 mg/dl. When blood glucose fell <180 mg/dl, insulin infusion will be tapered and eventually stopped. In the IGC group, insulin infusion will be started when blood glucose levels exceeded 140 mg/dl and adjusted to maintain glycemia at 80-140 mg/dl. During insulin infusion, oral feeding will be stopped and parenteral nutrition (13±5 Kcal/kg-1/day-1) will be started. After the start of insulin infusion protocol a glycemic control will be provided every hour in order to obtain three consecutive values that were within the goal range. The infusion will be lasted until stable glycemic goal (ICG group: 80-140 mg/dl; CGC group: 180-200 mg/dl) at least for 24 h. After glycemic goal will be maintained for 24 h, a parenteral nutrition was stopped and feeding will be started according to European guidelines. Subcutaneous insulin will be initiated at the cessation of the infusion. After discharge from the hospital, insulin will be given as short-acting insulin before meals and long-acting insulin in the evening for 30 days from PCI in both group. In IGC group, the treatment goal will be a fasting blood glucose level of 90-140 mg/dl and a non-fasting level of <180 mg/dl. In CGC group, the treatment goal will be fasting blood glucose and postprandial levels of <200 mg/dl. With regard to the full medical therapy, the protocol stated that the use of concomitant treatment should be as uniform as possible and according to evidence-based international guidelines for ACS. After 30 days from PCI, all patients with established diabetes and newly diagnosed diabetes will be managed and followed for 6 month after PCI, as outpatients, to maintain HbA1c <7% and blood glucose level of 90-140 mg/dl and a non-fasting level of <180 mg/dl.

Coronary Angiography Coronary angiograms at baseline, immediately after PCI, and at 6 months will be performed in at least 2 orthogonal views after intracoronary nitroglycerin. Minimum lumen diameter (MLD) and mean reference diameter (RD), obtained by averaging 5-mm segments proximal and distal to the target lesion location, will be used to calculate diameter stenosis as follows: (1-MLD/RD)X100. Late loss will the change in MLD from final PCI to follow-up. In-stent analysis will be confined to the stent itself, and in-segment analysis will be included the stent plus 5-mm segments proximal and distal to the stent. Binary restenosis will be defined as a <50% diameter stenosis. Qualitative analysis will be done with standard published methods.

IVUS Imaging and Analysis IVUS at baseline, immediately after PCI, and at 6 months will be performed with iLab, Galaxy, and ClearView or In Vision Gold with 20-MHz EagleEye catheters. IVUS imaging will be performed with motorized pullback at 0.5 mm/s to include the stent and >5 mm segments proximal and distal to the stent. IVUS studies will be archived onto super-VHS tape, CD-ROM, or DVD and will be sent to an independent, treatment-allocation- blinded, IVUS core laboratory for quantitative and qualitative analyses with validated planimetry software. Quantitative analysis will include measurement every 1 mm of the external elastic membrane (EEM), stent, and lumen cross-sectional areas (CSAs). Plaque plus media CSA will be calculated as EEM minus lumen. Neointimal hyperplasia (NIH) will be calculated as stent minus lumen. Once a complete set of CSA measurements will be obtained, intrastent and stent-edge volumes (EEM, plaque plus media, stent,lumen, and NIH) will be calculated with Simpson's rule and normalized for stent and reference segment length. Percent net volume obstruction will be calculated as NIH divided by stent volume.

Qualitative analysis will include stent malapposition (blood speckle behind stent struts), categorized as persistent (visible both at baseline and follow-up), resolved (visible only at baseline), and late acquired (only visible at follow-up); intrastent plaque and/or thrombus protrusion (IVUS cannot reliably differentiate between plaque and thrombus protruding through stent struts); stent fracture (absence of struts over more than one third of the stent circumference); aneurysm(lumen >50% larger than the proximal reference); and edge dissection.

ELIGIBILITY:
Inclusion Criteria:

* chest discomfort lasting at least 15 min within the last 24 h,
* new >l mm ST-wave or dynamic T-wave changes in at least two contiguous ECG leads,
* troponin I levels above the 99th percentile 6-12 h after the onset of chest pain
* patients referred to the cardiac catheterization laboratory within 24 h of symptoms.

Exclusion Criteria:

* left ventricular ejection fraction less than 25%,
* hemorrhagic diatheses,
* contraindications or allergy to aspirin, thienopyridines, and history of anaphylaxis in response to iodinated contrast medium,
* serum creatinine level of more than 2.0 mg/dl (177 μmol/l),
* leukocyte count of less than 3500/mm3, platelet count of less than 100,000/mm3
* coexisting conditions that limited life expectancy to less than 24 months or that could affect a patient's compliance with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Coronary angiograms | at baseline, immediately after PCI, and at 6 months

SECONDARY OUTCOMES:
IVUS Imaging | at baseline, immediately after PCI, and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Dept Geriatric and Metabolic diseases SUN, Naples, Italy, Italy

REFERENCES:
- [Derived] Marfella R, Rizzo MR, Siniscalchi M, Paolisso P, Barbieri M, Sardu C, Savinelli A, Angelico N, Del Gaudio S, Esposito N, Rambaldi PF, D'Onofrio N, Mansi L, Mauro C, Paolisso G, Balestrieri ML. Peri-procedural tight glycemic control during early percutaneous coronary intervention up-regulates endothelial progenitor cell level and differentiation during acute ST-elevation myocardial infarction: effects on myocardial salvage. Int J Cardiol. 2013 Oct 9;168(4):3954-62. doi: 10.1016/j.ijcard.2013.06.053. Epub 2013 Jul 19. PMID 23876463
- [Derived] Marfella R, Sasso FC, Siniscalchi M, Paolisso P, Rizzo MR, Ferraro F, Stabile E, Sorropago G, Calabro P, Carbonara O, Cinquegrana G, Piscione F, Ruocco A, D'Andrea D, Rapacciuolo A, Petronella P, Bresciani A, Rubino P, Mauro C, Paolisso G. Peri-procedural tight glycemic control during early percutaneous coronary intervention is associated with a lower rate of in-stent restenosis in patients with acute ST-elevation myocardial infarction. J Clin Endocrinol Metab. 2012 Aug;97(8):2862-71. doi: 10.1210/jc.2012-1364. Epub 2012 May 25. PMID 22639289